CLINICAL TRIAL: NCT06993935
Title: The Assessment of Health Literacy, Rational Drug Use, and Cyberchondria Levels in Individuals With Inflammatory Rheumatic Diseases
Brief Title: Health Literacy, Rational Drug Use, and Cyberchondria in Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Gülseren Demir Karakılıç, Assistant Professor, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 2024-GOKAEK-2411_2024.10.16_18
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis; Health Literacy; Rational Drug Use; Cyberchondria; Chronic Disease; Inflammatory Arthritis
Keywords: Rheumatic diseases, Knee osteoarthritis, Health literacy, Rational drug use, Cyberchondria
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Disease; Arthritis; Rheumatic Diseases; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient group: Patients who applied to the University Faculty of Medicine, Physical Medicine and Rehabilitation outpatient clinic, met the 2010 ACR criteria for Rheumatoid Arthritis, were aged 18 to 65, had intact cognitive functions, were literate, and consented to participate were included in the RA group; those who met the Modified New York criteria, were aged 18 to 65, had intact cognitive functions, were literate, and consented to participate were included in the AS group; and those who met the Classification of Psoriatic Arthritis (CASPAR criteria, were aged 18 to 65, had intact cognitive functions, were literate, and consented to participate were included in the PSA group
- Control patient group: After completing the surveys of patients with patient group, the gender and age distribution of the patient group was determined. The patient control group consisted of individuals who visited the Physical Medicine and Rehabilitation clinic of the University Faculty of Medicine due to knee pain lasting six months or longer, were diagnosed with knee osteoarthritis, matched the patient group in terms of age and gender, demonstrated adequate cognitive abilities, possessed literacy skills, and agreed to take part in the study.
- control group: The control group included healthy individuals who were of the same age and gender to the patient group, had good cognitive functions, were literate, had no disease or complaints, and agreed to take part in the study.

SUMMARY:
Purpose: This study aimed to evaluate rational drug use (RDU), health literacy (HL), and cyberchondria levels among individuals diagnosed with inflammatory rheumatic diseases, and to investigate the factors associated with these three key health-related variables.

Methods: This research was designed as a cross-sectional study and conducted between December 2024 and May 2025. The study enrolled three cohorts: a case cohort comprising patients diagnosed with rheumatic disease as patient group (group 1); a disease control cohort of knee osteoarthritis (group 2), and a reference control cohort of age- and sex-matched healthy participants (group 3). Disease Activity Score 28 (DAS28) was administered to patients with rheumatoid arthritis; Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) was administered to patients with ankylosing spondylitis; Psoriatic Arthritis Disease Activity Index (DAPSA) was administered to patients with psoriatic arthritis; Western Ontario and McMaster University Osteoarthritis Index (WOMAC) was administered to patients with knee osteoarthritis; and Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Turkey Health Literacy Scale-32 (THLS-32), Rational Drug Use Scale (RDUS), and Cyberchondria Severity Scale (CSS) were administered to all participants.

Results: The study sample consisted of 228 participants, with 76 individuals assigned to each of the three groups. Mean age, and gender distribution were similar in all three groups. Statistically significant variations were observed across the three groups regarding THLS-32, RDUS, and CSS scores (p < 0.001). Group 1 had the highest HL and RDUS scores, and moderate CSS scores. In contrast, Group 2 showed the lowest HL and RDUS scores, while Group 3 demonstrated the highest CSS scores. HL was positively correlated with RDU (r = 0.552, p < 0.001), and moderately negatively correlated with cyberchondria (r = -0.448, p < 0.001). These results indicate that higher HL is associated with more rational medication behavior and reduced susceptibility to online health-related anxiety. (p< 0.001).

Conclusions: To our knowledge, this is the first study to simultaneously investigate RDU and CSS in individuals diagnosed with RA, AS, and knee osteoarthritis. Our findings demonstrate that higher levels of HL are significantly associated with more appropriate medication behaviors and lower levels of internet-related health anxiety. These results emphasize the multidimensional role of HL, not only in promoting RDU but also in mitigating maladaptive digital health information-seeking patterns.

DETAILED DESCRIPTION:
Patient And Methods Study Design This prospective cross-sectional investigation was conducted from December 2024 to May 2025, involving both patient and control cohorts. Prior to enrollment, all participants provided written and verbal informed consent following a detailed explanation of the study objectives. The research protocol received full ethical approval from the Human Research Ethics Committee (2024-GOKAEK-2411_2024.10.16_188), ensuring adherence to international ethical guidelines. Patient enrollment start date: 22/12/2024, and ClinicalTrials.gov registration ID: NCT06348017.

Patients The study was commenced after obtaining the approval of the local ethics committee and the informed consent of the participants. Patients who applied to the University Faculty of Medicine, Physical Medicine and Rehabilitation outpatient clinic, met the 2010 ACR criteria for Rheumatoid Arthritis, were aged 18 to 65, had intact cognitive functions, were literate, and consented to participate were included in the RA group; those who met the Modified New York criteria, were aged 18 to 65, had intact cognitive functions, were literate, and consented to participate were included in the AS group; and those who met the Classification of Psoriatic Arthritis (CASPAR criteria, were aged 18 to 65, had intact cognitive functions, were literate, and consented to participate were included in the PSA group. After completing the surveys of patients with patient group, the gender and age distribution of the patient group was determined. The patient control group consisted of individuals who visited the Physical Medicine and Rehabilitation clinic of the University Faculty of Medicine due to knee pain lasting six months or longer, were diagnosed with knee osteoarthritis, matched the patient group in terms of age and gender, demonstrated adequate cognitive abilities, possessed literacy skills, and agreed to take part in the study. The control group included healthy individuals who were of the same age and gender to the patient group, had good cognitive functions, were literate, had no disease or complaints, and agreed to take part in the study.

The sociodemographic questionnaire, which was the data collection tool, was administered face-to-face to individuals at the Physical Medicine and Rehabilitation clinic along with several assessment scales: the Disease Activity Score 28 (DAS28), the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), the Disease Activity Index for Psoriatic Arthritis (DAPSA), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the Beck Depression Inventory (BDI), and the Beck Anxiety Inventory (BAI), as well as the Turkey Health Literacy Scale-32 (THLS-32), the Rational Drug Use Scale (RDUS), and the Cyberchondria Severity Scale (CSS).

DAS28: In patients with RA, disease activity is assessed using the DAS28 scale. This method is a widely used tool to determine disease activity in RA. The evaluation involves assessing 28 joints for tenderness and swelling. The patient's global pain assessment score, along with C-reactive protein (CRP) levels or erythrocyte sedimentation rate (ESR), is entered into a computer program to calculate the DAS28 score. A total score >5.1 indicates high disease activity, a score between 3.2-5.1 indicates moderate disease activity, a score <3.2 indicates low disease activity, and a score <2.6 is considered remission [29].

BASDAI: The BASDAI is used to evaluate disease activity in patients with AS. As the BASDAI score increases, the level of disability associated with the disease also rises. A BASDAI score ≥4 indicates active disease. The Turkish validity and reliability study of the BASDAI was conducted in 2005 [30].

DAPSA: Disease activity in patients with PSA is assessed using the DAPSA score. This method is based on the evaluation of 68 joints for tenderness and 66 joints for swelling. The number of tender and swollen joints, the pain assessment score via the Visual Analog Scale (VAS), the physician's global assessment, and CRP values are summed to calculate the DAPSA score. A score >28 indicates high disease activity, a score between 15-28 indicates moderate disease activity, a score between 5-14 indicates low disease activity, and a score <4 is considered remission [31].

WOMAC: is a tool commonly used to assess the level of functional impairment in patients with knee osteoarthritis. It includes 24 items divided into three domains: pain, stiffness, and physical function. Each item is rated on a scale from 0 (none) to 4 (extreme), with higher total scores reflecting greater severity of symptoms and functional limitations. The Turkish adaptation of the WOMAC was validated by Tüzün et al. [32].

BDI: is developed by Beck and colleagues in 1961, is intended to evaluate the typical signs and symptoms associated with depression. This instrument is a self-administered questionnaire comprising 21 items and usually requires around 10 minutes to complete. The Turkish version of the inventory was adapted and validated by Hisli and colleagues [33].

BAI: is developed by Aaron T. Beck, is an internationally validated tool for assessing anxiety levels. It consists of 21 items. The Turkish adaptation and validation of the inventory were performed by Ulusoy and colleagues [34].

THLS-32: Developed and validated by Okyay and colleagues [35], the THLS-32 measures HL levels. It has two sub-groups: treatment service score and disease prevention score, but there is no separate cut-off value determined for these sub-scales; the higher the score, the higher the literacy. Scores range from 0 to 50, where 0 indicates the lowest and 50 the highest level of HL. HL levels are categorized as follows: 0-25 points indicate "inadequate" HL, >25-33 points indicate "problematic/limited," >33-42 points indicate "adequate," and >42-50 points indicate "excellent" HL.

RDUS: Developed by Demirtaş and colleagues, this scale has undergone a Turkish validity and reliability study [36]. It consists of 21 items scored on a 3-point Likert scale. Responses are scored as "correct answer = 2 points," "I don't know = 1 point," and "wrong answer = 0 points." Total scores range from 0 to 42, with higher scores indicating better levels of RDU. A cutoff score of 34 and above is interpreted as "good RDU." The Cronbach's alpha coefficient for the scale is 0.78.

CSS: Adapted into Turkish by Uzun and Zencir [37], this scale comprises 33 items rated on a 5-point Likert scale, ranging from "Never" to "Always." The scale has five subdimensions: compulsion, excessive concern, excessive searching, reassurance seeking, and distrust of medical professionals. Compulsion, excessive concern, and excessive searching subscales range from 8 to 40 points, reassurance seeking ranges from 6 to 30 points, and distrust of medical professionals ranges from 3 to 15 points. The total score ranges from 33 to 165, with higher scores indicating higher levels of cyberchondria. The overall Cronbach's alpha coefficient of the scale is 0.94.

Statistical analysis Sample analysis was performed using the Openepi application https://www.openepi.com/SampleSize/SSPropor.htm). Based on the study by Kalmaz et al., it was determined that at least 75 participants should be included in each group for a margin of error of 0.05, an effect size of 0.465, and 95% power [28]. Data analysis was conducted using SPSS version 25.0 (SPSS Inc., Armonk, NY). The Kolmogorov-Smirnov test was applied to assess the normality of continuous variables. Categorical data were evaluated with Pearson's Chi-Square Test or Fisher's Exact Test depending on the expected frequencies. For continuous variables, group differences were analyzed using the Student's T-Test or One-Way Analysis of Variance (ANOVA). When multiple group comparisons were necessary, post-hoc analyses were performed using Tukey's or Games-Howell tests. Spearman's correlation coefficients were calculated to explore relationships between variables and disease activity or scale scores, including DAS28, BASDAI, DAPSA, WOMAC, BDI, BAI, THLS-32, RDUS, and CSS within the patient cohort.

ELIGIBILITY:
Inclusion Criteria:

Obtained approval from the local ethics committee. Provided informed consent to participate. Aged 18 to 65 years. Possessed intact cognitive functions. Literate. For the Rheumatoid Arthritis (RA) group: Met the 2010 ACR criteria for Rheumatoid Arthritis.

For the Ankylosing Spondylitis (AS) group: Met the Modified New York criteria. For the Psoriatic Arthritis (PsA) group: Met the Classification of Psoriatic Arthritis (CASPAR) criteria.

For the Knee Osteoarthritis (KOA) control group:

Visited the Physical Medicine and Rehabilitation clinic due to knee pain lasting six months or longer.

Diagnosed with knee osteoarthritis. Matched the patient group in terms of age and gender. Demonstrated adequate cognitive abilities. Possessed literacy skills.

For the Healthy control group:

Same age and gender as the patient group. Had good cognitive functions. Literate. Had no disease or complaints.

Exclusion Criteria:

Under the age of 18 or over the age of 65. Any condition that could impair communication. Refusal to participate in the study. Not possessing digital devices such as a smartphone or computer, or lacking internet access.

Illiterate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adults aged 18 to 65 years, including patients diagnosed with rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, or knee osteoarthritis, as well as healthy controls matched for age and gender. All participants had sufficient cognitive abilities, were literate, and consented to participate.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Turkey Health Literacy Scale-32 (THLS-32) | At enrollment
  Developed and validated by Okyay and colleagues, the THLS-32 measures HL levels. It has two sub-groups: treatment service score and disease prevention score, but there is no separate cut-off value determined for these sub-scales; the higher the score, the higher the literacy. Scores range from 0 to 50, where 0 indicates the lowest and 50 the highest level of HL. HL levels are categorized as follows: 0-25 points indicate "inadequate" HL, >25-33 points indicate "problematic/limited," >33-42 points indicate "adequate," and >42-50 points indicate "excellent" HL.
Rational Drug Use Scale (RDUS), | At enrollment
  Developed by Demirtaş and colleagues, this scale has undergone a Turkish validity and reliability study. It consists of 21 items scored on a 3-point Likert scale. Responses are scored as "correct answer = 2 points," "I don't know = 1 point," and "wrong answer = 0 points." Total scores range from 0 to 42, with higher scores indicating better levels of RDU. A cutoff score of 34 and above is interpreted as "good RDU." The Cronbach's alpha coefficient for the scale is 0.78.
Cyberchondria Severity Scale (CSS) | At enrollment
  Adapted into Turkish by Uzun and Zencir, this scale comprises 33 items rated on a 5-point Likert scale, ranging from "Never" to "Always." The scale has five subdimensions: compulsion, excessive concern, excessive searching, reassurance seeking, and distrust of medical professionals. Compulsion, excessive concern, and excessive searching subscales range from 8 to 40 points, reassurance seeking ranges from 6 to 30 points, and distrust of medical professionals ranges from 3 to 15 points. The total score ranges from 33 to 165, with higher scores indicating higher levels of cyberchondria. The overall Cronbach's alpha coefficient of the scale is 0.94.
the Disease Activity Score 28 (DAS28) | At enrollment
  In patients with RA, disease activity is assessed using the DAS28 scale. This method is a widely used tool to determine disease activity in RA. The evaluation involves assessing 28 joints for tenderness and swelling. The patient's global pain assessment score, along with C-reactive protein (CRP) levels or erythrocyte sedimentation rate (ESR), is entered into a computer program to calculate the DAS28 score. A total score >5.1 indicates high disease activity, a score between 3.2-5.1 indicates moderate disease activity, a score <3.2 indicates low disease activity, and a score <2.6 is considered remission.
the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), | At enrollment
  The BASDAI is used to evaluate disease activity in patients with AS. As the BASDAI score increases, the level of disability associated with the disease also rises. A BASDAI score ≥4 indicates active disease. The Turkish validity and reliability study of the BASDAI was conducted in 2005.
the Disease Activity Index for Psoriatic Arthritis (DAPSA) | At enrollment
  Disease activity in patients with PSA is assessed using the DAPSA score. This method is based on the evaluation of 68 joints for tenderness and 66 joints for swelling. The number of tender and swollen joints, the pain assessment score via the Visual Analog Scale (VAS), the physician's global assessment, and CRP values are summed to calculate the DAPSA score. A score >28 indicates high disease activity, a score between 15-28 indicates moderate disease activity, a score between 5-14 indicates low disease activity, and a score <4 is considered remission.
the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), | At enrollment
  is a tool commonly used to assess the level of functional impairment in patients with knee osteoarthritis. It includes 24 items divided into three domains: pain, stiffness, and physical function. Each item is rated on a scale from 0 (none) to 4 (extreme), with higher total scores reflecting greater severity of symptoms and functional limitations. The Turkish adaptation of the WOMAC was validated by Tüzün et al.
the Beck Depression Inventory (BDI), | At enrollment
  BDI: is developed by Beck and colleagues in 1961, is intended to evaluate the typical signs and symptoms associated with depression. This instrument is a self-administered questionnaire comprising 21 items and usually requires around 10 minutes to complete. The Turkish version of the inventory was adapted and validated by Hisli and colleagues.
the Beck Anxiety Inventory (BAI), | At enrollment
  is developed by Aaron T. Beck, is an internationally validated tool for assessing anxiety levels. It consists of 21 items. The Turkish adaptation and validation of the inventory were performed by Ulusoy and colleagues.
Visual Analog Scale (VAS) | At enrollment
  For the Evaluation of Pain. For this evaluation, the patient is asked to mark their pain and fatigue severity on a horizontal 10-cm line with the number 0 on one end representing "no pain or no fatigue" and the number 10 on the other end indicating "very severe pain or very severe fatigue."

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Asst Prof, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months after study completion

REFERENCES:
- [Background] Akkoc Y, Karatepe AG, Akar S, Kirazli Y, Akkoc N. A Turkish version of the Bath Ankylosing Spondylitis Disease Activity Index: reliability and validity. Rheumatol Int. 2005 May;25(4):280-4. doi: 10.1007/s00296-003-0432-y. Epub 2004 Jan 17. PMID 14730386